CLINICAL TRIAL: NCT01517139
Title: Pilot Study to Test the Methods for the Diet, Nutrition and Physical Activity Feasibility Study of Early Life Determinants of Adult Cancers in a Chinese Cohort of Adolescents and Their Mothers
Brief Title: Diet and Nutrition Pilot Study for Chinese Adolescents and Their Mothers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912038; 12-C-N038
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Methylation; Body Composition; Physical Activity; Puberty
Keywords: Diet and Nutrition; Pregnancy Folic Acid; In Utero Exposure; DNA Methylation; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Feasibility Cohort: 100 pairs of children and their mothers recruited from 2 provinces.

SUMMARY:
Background:

- Researchers want to collect information on diet, physical activity, and sun exposure in children and young adults. The data can provide information on the effect these factors might have on the development of cancer and other diseases. Information collected only from adults does not accurately measure these factors. To collect more accurate information, both mothers and children will provide information. Study participants will be from Hebei province in northeastern China and Jiangsu province in eastern China.

Objectives:

- To collect and study diet, activity, and sun exposure data from Chinese adolescents and their mothers.

Eligibility:

* Adolescents between 15 and 17 years of age from Hebei and Jiangsu provinces in China.
* Mothers of the study adolescents.

Design:

* Participants will answer questions about their diet, physical activity, and time in the sun.
* Participants will wear a pedometer to measure activity for 7 days. They will also wear a badge to measure sun exposure for 3 days.
* Participants will record their activities and food and drinks consumed for 3 days. Urine samples will be collected for a full day.
* Participants will have a grip strength test. On the last day of the study, they will provide blood, saliva, and toenail samples.
* A smaller separate group of adolescents will provide saliva samples only and complete a food questionnaire.

DETAILED DESCRIPTION:
Background:

Emerging epidemiological evidence suggests that early-life exposures in conjunction with genetic makeup and variability may be important in the etiology of many common adult cancers. Prospectively collected information on adolescent and early adulthood exposures is lacking and current evidence often relies on adult recall of the past with a limited array of exposure variables.

Long Term Objective:

1. To investigate the feasibility of assessing exposures that may be linked to early life exposures and to later diseases. Exposures include diet, physical activity, UV-exposure, DNAmethylation status, body size and reproductive factors. This feasibility work will inform additional research in an existing large Chinese-U.S. CDC collaborative project conducted in 1993 - 1995, the Community Intervention Program (CIP) (n = 247,000).

   Short Term Objectives:
2. To determine the feasibility of collecting and assessing the quality of data on current diet, nutritional status, physical activity, physical strength, UV exposure, DNA methylation status and other environmental exposures as early life determinants of adult cancer in adolescents 15 - 17 years of age and early adulthood in their mothers.
3. To assess differences in methylation status of DNA between those exposed to periconceptional folic acid supplementation and those unexposed.
4. To compare dietary and physical activity self-reporting instruments against objective measures of dietary intake and physical activity, respectively.

Eligibility:

Pairs of mothers and their children aged 15-17 years from the CIP, who completed an associated pilot study in Laoting (Task 1), Hebei provincein the North, and Taicang, Jiangsu provincein the South, and who agree to participate in the study. An additional subsample of 100 children who completed an accompanying study (Task 1), who agree to participate in a sub-study will be eligible.

Design:

This pilot study will include 100 pairs of children and their mothers recruited from 2 provinces. A total of 50 children (aged 16-17years) from a high school (grades 9-10) will be identified in each province. To the extent possible, approximately equal numbers of children aged 16 and 17 years of age will be recruited, stratified by gender and in utero exposure to folic acid. An additional sub-sample of 100 children that completed an accompanying study (Task 1) will be enrolled for only saliva collection and completion of a food frequency questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pairs of mothers and their children 15 - 17 years of age who completed Task1 and who agree to participate in the study (Task2 ).

EXCLUSION CRITERIA:

1. Maternal pill usage only after conception and those who may have stopped taking folic acid pills before the second trimester.
2. Pairs of mothers and children where the mother is not the primary guardian (e.g., mother died or never lived with the child).

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a pilot study of approximately 200 children and their mothers who had participated in a prior study of 247,000 mother-child pairs in 1993 to 1995. The aim of the pilot is to assess the feasibility of finding the subjects, assessing participation rates, and testing instruments to measure diet, physical activity and ultraviolet radiation exposure. Participants were identified from records documenting location of residence in the previous study. They were approached by local medical staff to assess interest in participation for the pilot study. The study involved 8 days of data collection as well as saliva and blood collection. Results from the local hospital blood tests and the research sample were provided to the participants by the local medical staff. Follow-up of the larger cohort would be based on successful study protocol components or improved versions of the instruments or logistics.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2013-08-27 (Actual)

PRIMARY OUTCOMES:
Participation rates >60% | At the end of the study, July 2012
  Participation rates were 66% in the rural community and 87% in the urban community.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Potischman, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Chinese Center for Disease Contron & Prevention, Beijing, China